CLINICAL TRIAL: NCT07373899
Title: Comparison of the Effect of Surgical Resection Based on Lesion Extent Before and After Neoadjuvant Therapy in Patients With Stage II-IIIB Non-Small Cell Lung Cancer: A Single-Center, Real-World, Open-Label Study
Status: Not yet recruiting | Type: Observational
Sponsor: Cancer Institute and Hospital, Chinese Academy of Medical Sciences (Other)
Responsible Party: Sponsor
Other Study IDs: NCC5959
Record Dates: First submitted 2026-01-20; First posted 2026-01-28 (Actual); Last update posted 2026-01-28 (Actual); Status verified 2025-12

CONDITIONS: Carcinoma, Non-Small-Cell Lung; Neoadjuvant Immunotherapy; Surgery
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Conventional Surgery Group: Perform a pneumonectomy or composite lobectomy within the originally planned scope
- Modified/Reduced Surgery Group: Under the premise of ensuring R0 resection, reduce the surgical scope, prefer composite lobectomy or lobectomy to maximize the preservation of pulmonary function.

SUMMARY:
This study intends to conduct a prospective, non-interventional study to compare the survival benefits of different surgical resection patterns for patients with non-small cell lung cancer who have achieved partial response (PR) after immunotherapy induction. The study plans to enroll patients suitable for surgery as assessed by radiomics evaluation and multidisciplinary team (MDT) discussion, and will assign them to the modified surgery group and the conventional surgery group based on patient preference. The resection scope in the modified surgery group is more limited compared to conventional surgery, aiming to maximize preservation of pulmonary function while ensuring oncological safety. This study will systematically evaluate the impact of different resection scopes on patient prognosis after neoadjuvant immunotherapy, providing clinical evidence for exploring individualized surgical strategies for non-small cell lung cancer in the era of immunotherapy.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed NSCLC; ② Achieved resectable criteria after neoadjuvant immunotherapy (± chemotherapy); ③ Originally required total lung resection or combined lobectomy based on the size and extent of the lesion, but after neoadjuvant treatment, the condition was suitable for minimally invasive resection; ④ Age ≥ 18 years; ⑤ ECOG score 0-1; ⑥ Complete imaging, pathological and follow-up data.

Exclusion Criteria:

* ① Disease progression (PD) after neoadjuvant therapy; ② Those who still require total lung resection or combined lobectomy and whose scope cannot be reduced; ③ During the operation, it is found that R0 resection is impossible; ④ Severe cardiopulmonary dysfunction or other complications make them intolerant to surgery.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All the patients were those admitted to the Thoracic Surgery Department of the Cancer Hospital of Chinese Academy of Medical Sciences.
Sampling Method: Non-Probability Sample
Enrollment: 354 (Estimated)
Dates: Start 2026-01-01 (Estimated); Primary Completion 2030-12-31 (Estimated); Study Completion 2030-12-31 (Estimated)

PRIMARY OUTCOMES:
Disease-free survival | Evaluate over a period of up to five years
  It refers to the period from the beginning of the study until the recurrence of the disease or any cause of death.

SECONDARY OUTCOMES:
Overall Survival (OS) | From date of diagnosis until the date of death from any cause, whichever came first, assessed up to 5 years.
  OS is defined as the time from surgery time until death from any cause.
Pathological Complete Response(pCR) | up to 1 month after surgery
  After evaluating the removed tumor tissue and the regional lymph nodes, no residual tumor cells were found.
Incidence of perioperative complications | up to 1 month after surgery
  The perioperative period refers to a certain period before, during and after the surgery. Postoperative pulmonary complications refer to various respiratory system complications that occur in patients after the surgery.